CLINICAL TRIAL: NCT00657085
Title: Evaluation of the LightSheer HS Hand Piece as Compared to the LightSheer ET Hand Piece for the Intended Use of Hair Removal and Permanent Hair Reduction
Status: Completed | Type: Observational
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Chris Clark, Lumenis
Other Study IDs: LUM-ABU-HSET-0607-02
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Laser Hair Removal
Keywords: Laser hair removal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsied hair follicles retained and analzed through horizontal sectioning and viability staining
Oversight: Data Monitoring Committee: No

SUMMARY:
To observe the qualitative comparison of follicular damage between treatment with the LightSheer Duet hand pieces (ET and HS) as assessed by horizontal biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adult, 18 years of age or older with skin type I-V;
2. Having a suitable treatment area for hair removal with brown or black hair (no gray);
3. Able and willing to comply with the treatment/follow-up schedule and requirements;
4. Able to read, understand and provide written Informed Consent.

Exclusion Criteria:

1. Showing symptoms of hormonal disorders, as per the Investigator's discretion;
2. Use of oral isotretinoin (Accutane®) within 6 months, or off label use of topical isotretinoin in immediate treated area or in its proximity within 3 months, of study enrollment or during the course of the study;
3. Prior skin treatment with laser or other devices on the same treated areas prior to study enrollment or during the course of the study;
4. Adverse reaction to the treatment gel to be used in the evaluation;
5. History of keloid formation or poor wound healing in a previously injured skin area;
6. Significant skin conditions affecting treated area or inflammatory skin conditions;
7. Open laceration, abrasion, active cold sores or herpes sores on area to be treated;
8. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications;
9. Having a bleeding disorder or taking anticoagulation medications within the preceding 6 months;
10. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the area to be treated;
11. Significant concurrent illness, such as diabetes, lupus, epilepsy or cardiac disorders, which might be aggravated as a result of treatment;
12. Unable or unlikely to refrain from tanning, including the use of tanning booths, tanning spray or cream, during the course of the evaluation;
13. Photosensitivity disorder that can be exacerbated by infrared light;
14. Tattoos in the treatment areas;
15. Dysplastic nevi in the treatment areas;
16. Allergy or history of an allergy to the topical anesthetic used.
17. Participation in a study of another device or drug within 3 months prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria;
18. Mentally incompetent, prisoner or evidence of active substance or alcohol abuse;
19. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 5 Adult male subjects that have sought laser back hair removal
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Follicular damage assessed by histology | first visit

SECONDARY OUTCOMES:
Comparison of permanent hair reduction between ET and HS handpieces | 2 month follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Seaver Soon, MD, Principal Investigator — Scripps Dermatology
Locations (1):
- Seaver Soon, San Diego, California, United States